CLINICAL TRIAL: NCT01119287
Title: A Randomized, Double-Masked, Placebo-Controlled, Parallel Group Study to Assess the Efficacy of Maxidex® (0.1% Dexamethasone) Ophthalmic Suspension and Patanol® (0.1% Olopatadine Hydrochloride) Ophthalmic Solution for the Treatment of Allergic Conjunctivitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: Assessing the Efficacy of Maxidex® and Patanol® for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: C-10-002
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2013-03

CONDITIONS: Allergic Conjunctivitis
Keywords: Conjunctivitis; ocular allergy
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — Dexamethasone; Olopatadine Hydrochloride; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maxidex (Experimental): Dexamethasone 0.1% ophthalmic suspension, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
  Interventions: Drug: Dexamethasone 0.1% ophthalmic suspension
- Patanol (Experimental): Olopatadine hydrochloride 0.1% ophthalmic solution, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
  Interventions: Drug: Olopatadine hydrochloride 0.1% ophthalmic solution
- Tears Naturale II (Placebo Comparator): Inactive ingredients, used as placebo, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
  Interventions: Other: Inactive ingredients, used as placebo

INTERVENTIONS:
Drug: Dexamethasone 0.1% ophthalmic suspension — Maxidex
  Arms: Maxidex
Drug: Olopatadine hydrochloride 0.1% ophthalmic solution — Patanol
  Arms: Patanol
Other: Inactive ingredients, used as placebo — Tears Naturale II
  Arms: Tears Naturale II

SUMMARY:
The purpose of this study was to evaluate the efficacy of Maxidex and Patanol compared to placebo in patients with allergic conjunctivitis when exposed to controlled allergen levels in an Environmental Exposure Chamber (EEC).

DETAILED DESCRIPTION:
This study consisted of 6 visits. Visit 1 was the Medical Screening Visit (skin prick test). Visit 2 and Visit 3 consisted of 2 consecutive EEC Visits (3 hours in the EEC followed by 7 hours in the Clinic, 10 hours total, each visit) followed by 7 days of wash-out. Visit 2 and Visit 3 occurred prior to dispense and the measures obtained during these visits were used as baseline. At Visit 4 patients were randomized and dispensed the assigned study medication for 7 days of at-home dosing. Visit 5 (Day 8 of treatment) and Visit 6 (Day 9 of treatment) consisted of 2 additional consecutive EEC Visits (3 hours in the EEC followed by 7 hours in the clinic, 10 hours total, each visit). During each EEC visit, patients were exposed to either ragweed or cat allergen, depending on their skin prick test results. Of the 180 participants enrolled, 170 received at least one dose of study treatment and were randomized to one of the three study treatments.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year history of allergic conjunctivitis.
* Ability to self administer ophthalmic drops.
* Ability to avoid use of disallowed medications during the entire study period and specified period prior to visit 1.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Presence of any ocular infection.
* Confirmed diagnosis of dry eye.
* Presence of glaucoma or ocular hypertension.
* Moderate to severe asthma.
* Any severe, unstable, or uncontrolled systemic disease.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from one study center in Canada.
Pre-assignment Details: Of the 180 patients enrolled, 170 were identified as either ragweed allergic or cat allergic, randomized to one of three study treatments, and received at least one dose of study treatment. Ten additional patients identified as ragweed allergic participated in Visits 1 to 3 only, per protocol design.
Groups:
- Maxidex/Ragweed Allergic; Maxidex/Cat Allergic: Dexamethasone 0.1% ophthalmic suspension, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
- Patanol/Ragweed Allergic; Patanol/Cat Allergic: Olopatadine hydrochloride 0.1% ophthalmic solution, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
- Tears Naturale II/Ragweed Allergic; Tears Naturale II/Cat Allergic: Inactive ingredients, used as placebo, 2 drops in each eye, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
Period: Overall Study
Arm/Group | Maxidex/Ragweed Allergic | Patanol/Ragweed Allergic | Tears Naturale II/Ragweed Allergic | Maxidex/Cat Allergic | Patanol/Cat Allergic | Tears Naturale II/Cat Allergic
Started | 26 | 24 | 26 | 31 | 31 | 32
Completed | 26 | 24 | 24 | 29 | 30 | 32
Not Completed | 0 | 0 | 2 | 2 | 1 | 0
Not completed — Patient Decision, not related to AE | 0 | 0 | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maxidex/Ragweed Allergic | Patanol/Ragweed Allergic | Tears Naturale II/Ragweed Allergic | Maxidex/Cat Allergic | Patanol/Cat Allergic | Tears Naturale II/Cat Allergic | Total
Number analyzed (Participants) | 26 | 24 | 26 | 31 | 31 | 32 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.6) | 39.2 (13.8) | 40.0 (10.0) | 34.5 (11.6) | 32.9 (9.3) | 35.9 (8.4) | 35.91 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 17 | 23 | 22 | 24 | 110
  Male | 15 | 11 | 9 | 8 | 9 | 8 | 60
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 24 | 26 | 31 | 31 | 32 | 170

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Staff-Assessed Ocular Redness, Area Under the Curve From Time Zero to Hour 10 [AUC (0-10)], Maxidex and Placebo
Description: Ocular redness ratings were collected for nasal and temporal areas of each eye and scored on a scale from 0 (none) to 4 (extremely severe), 0.5 unit steps permitted. The AUC computation was based on peak redness score (maximum of four areas of redness) at each time point (pre-treatment, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3 hours in the EEC and 3.5, 4, 5, 6, 7, 8, 9, 10 hours in the Clinic). The patient was dosed AM 30 minutes prior to entering the EEC (Visit 6). This outcome measure evaluates a late-phase effect, for which Maxidex vs. Placebo is the meaningful comparison.
Time Frame: Baseline (Visit 3, pre-treatment); Visit 6 (Day 9 of treatment)
Population: Number of subjects with data available in the specific treatment group
Measure: Mean (Standard Deviation); unit: hours x units on a scale
Arm/Group | Maxidex/Ragweed Allergic | Tears Naturale II/Ragweed Allergic | Maxidex/Cat Allergic | Tears Naturale II/Cat Allergic
Number analyzed (Participants) | 26 | 24 | 29 | 32
hours x units on a scale
  Baseline (Visit 3, pre-treatment) | 18.120 (6.260) | 19.362 (7.666) | 16.823 (5.530) | 17.572 (6.803)
  Visit 6 (Day 9 of treatment) | 11.671 (5.983) | 15.786 (6.514) | 11.313 (3.943) | 13.824 (4.792)
  Change | -6.450 (7.002) | -3.576 (6.959) | -5.511 (5.916) | -3.748 (6.351)

2. Primary Outcome: Mean Change From Baseline Patient-Assessed Ocular Itching, Area Under the Curve From Time Zero to Hour 3 [AUC (0-3)], Patanol and Placebo
Description: Ocular itching was scored a scale from 0 (none) to 4 (incapacitating itch with irresistible urge to rub) in 0.5 unit steps. The AUC computation was based on the score at each time point (pre-treatment, 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, and 3 hours in the EEC). The patient was dosed AM 30 minutes prior to entering the EEC (Visit 5). This outcome measure evaluates an early-phase effect, for which Patanol vs. Placebo is the meaningful comparison.
Time Frame: Baseline (Visit 2, pre-treatment), Visit 5 (Day 8 of treatment)
Population: Number of subjects with data available in the specific treatment group
Measure: Mean (Standard Deviation); unit: hours x units on a scale
Groups:
- Tears Naturale II/Ragweed Allergic: Inactive ingredients, used as placebo, 2-5 minutes apart, twice a day, for 9 days [Visit 4 through Visit 6 morning only]
Arm/Group | Patanol/Ragweed Allergic | Tears Naturale II/Ragweed Allergic | Patanol/Cat Allergic | Tears Naturale II/Cat Allergic
Number analyzed (Participants) | 24 | 24 | 30 | 32
hours x units on a scale
  Baseline (Visit 2, pre-treatment) | 4.776 (1.759) | 5.669 (2.062) | 5.904 (2.224) | 5.654 (2.408)
  Visit 5 (Day 8 of treatment) | 2.630 (1.877) | 3.990 (2.781) | 2.881 (2.203) | 2.586 (2.181)
  Change | -2.146 (1.913) | -1.680 (2.065) | -3.023 (2.668) | -3.068 (2.361)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (5 months, 29 days).
Description: The safety population included all randomized patients. Adverse events were reported for any clinically relevant untoward (unfavorable and unintended) change from baseline in the patient's medical health following exposure to the study treatment, as reported spontaneously by the patient and solicited by the investigator.
Arm/Group | Maxidex | Patanol | Tears Naturale II
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/55 | 0/58
Other Adverse Events (participants affected / at risk) | 13/57 | 7/55 | 7/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maxidex (N=57) | Patanol (N=55) | Tears Naturale II (N=58)
Eye irritation (Eye disorders) | 4 | 4 | 4
Eye pain (Eye disorders) | 5 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other